CLINICAL TRIAL: NCT02217306
Title: Contrast Sensitivity and Diabetic Macular Edema
Status: Completed | Type: Observational
Sponsor: Hospital Juarez de Mexico (Other Government)
Responsible Party: Principal Investigator, Dulce Milagros Razo Blanco Hernández, MEDICAL RESEARCHER, Hospital Juarez de Mexico
Other Study IDs: HJM2295/14R
Record Dates: First submitted 2014-08-06; First posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: DIABETES MELLITUS; DIABETIC RETINOPATHY; MACULAR EDEMA
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy; Macular Edema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Contrast Sensitivity: Determine changes in contrast sensitivity frequences and visual function (visual acuity) after one month of treatment photocoagulation in macular edema

SUMMARY:
Contrast sensitivity is a tool use to evaluate the visual function in all patients. It can be modified by different pathologies or by age. The purpose of this study is to identify the changes that could be in relationship with the course of diabetic retinopathy comparing with diabetic patient without retinopathy and in patients with diabetic macular edema so if it is a difference, research for therapeutic strategies to improve it in this patients.

DETAILED DESCRIPTION:
Contrast sensitivity is defined as a subjective measurement, it is the ability to separate the image between figure and background, taking into account the minimum amount of light required; it is evaluated by the contrast threshold, which is the smallest amount of contrast needed to be able to see a target and solve their characteristics, would be his reciprocal value. Medina et al. curve reported in healthy Mexicans SC 5 to 80, where > 51 years have decreased compared to contrast sensitivity studies international; further that contrast sensitivity in older groups of 41 years is decreased high frequency.

ELIGIBILITY:
Inclusion Criteria:

* DIABETIC PATIENTS
* 40-60 YEARS OLD
* ANY GENDER
* VISUAL ACUITY >0.25 IN DECIMAL EQUIVALENT,

Exclusion Criteria:

* PATIENTS WITH CATARACTS OR OTHER MACULOPATHY
* PATIENTS WITH CONTACT LENSES
* PATIENTS WITH REFRACTIVE ERROR >6.00DP
* PATIENTS WITH PREVIOUS OCULAR SURGERY

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients attended at Ophthalmology service in a general hospital
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Contrast Sensitivity | up to 8 months
  Diabetic patients who are attended at Ophthalmology service in a general hospital undergo to contrast sensitivity test evaluating all frequency by software with 5 spacial frequency (1.5, 3, 6, 12 and 18 cycle grade, Stereoptical Co 1996) in the Visual Basic program.

CONTACTS AND LOCATIONS:
Overall Officials: DULCE MI RAZO BLANCO HERNANDEZ, MD, Principal Investigator — Hospital Juarez de Mexico; SURISADAI SERAFIN SOLIS, MSc, Study Chair — INSTITUTO POLITECNICO NACIONAL; LOURDES CA ORTEGA LUNA, MSc, Study Chair — INSTITUTO POLITECNICO NACIONAL; VIRGILIO LIMA GOMEZ, MD, MSc, Study Director — Hospital Juarez de Mexico
Locations (1):
- Hospital Juarez de Mexico, Mexico City, Mexico City, Mexico